CLINICAL TRIAL: NCT04136561
Title: Novel Strategy to Encourage Early Removal of Central Venous Catheters
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled. Unable to enroll
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Amit Bahl, Director Emergency Medicine Ultrasound, Corewell Health East
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-235
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Vascular Access Complication; Central Line Complication; Central Line-Associated Infection; Superficial Vein Thrombosis; Deep Vein Thrombosis
Keywords: intravenous access; vascular access; IV survival; IV catheter complication; Central venous access; Central Line-associated Bloodstream Infection (CLABSI)
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Prospective with historical case matched controls, Non-randomized, Single site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CVC and Midline Catheter (Experimental): Existing standard of care CVC. Midline catheter placed within 24 hours of CVC placement.
  Interventions: Device: Midline catheter
- CVC (No Intervention): Standard of care CVC: case-matched controls using baseline data.

INTERVENTIONS:
Device: Midline catheter — Midline catheter placed in patients with existing standard of care CVC
  Arms: CVC and Midline Catheter

SUMMARY:
The goal of this study is to determine if early placement of a midline catheter in patients with a central venous catheter (CVC) will decrease the number of days the CVC is in place. Patients who are in the medical intensive care unit (MICU) and have a CVC may be approached to join the study. Those who meet study eligibility and provide written consent will be enrolled. The longer the CVC remains in place,the greater the chance of developing an infection or blood clot. Any IV line that is placed (CVC, midline, peripheral line) comes with the risk of infection or blood clots, although that risk is generally less with the midline and peripheral IV lines than a CVC. The treating team will make the decision when to remove the CVC. The timeline of removal will be compared to previous data collected on patients similar to the ones in this study. During their hospital stay, study patients will be monitored for how well the midline catheter is functioning as well as if they develop a catheter related blood clot or infection.

DETAILED DESCRIPTION:
Central line-associated bloodstream infection (CLABSI) remains a serious problem contributing to patient morbidity and mortality. These potentially preventable complications have high costs. Significant interventions focusing on insertion of catheter and care and maintenance protocols have been helpful in reducing CLABSI rates. One component that remains a challenge is early/appropriate removal of central venous catheters (CVCs). The longer the central line remains in the patient, the increased chance of developing a CLABSI.

The study design is case-controlled with a control group composed of patients admitted in the previous year who received a CVC as part of the treatment plan and who did not received a midline catheter.The intervention phase of this study will involve placement of a standard of care, FDA approved midline catheter in patients that have a CVC. The Medical Intensive Care Unit (MICU) treating team will be consulted prior to approaching the patient. Written informed consent will be obtained from the patient or legal authorized representative prior to enrollment. The midline catheters will be inserted by the vascular access team within 24 hours of CVC insertion. Midline catheters will be assessed daily for function, phlebitis, and infection for up to 7 days. Mechanical complications or premature line failures will be tracked. Data specific to blood sampling will be collected daily. If the catheter was identified to have failed during follow-up assessment the date and time of failure and the reason for failure will be documented. If the catheter failed or was removed prior to the follow-up assessment then the VAD failure time and the assessment of failure and reason for line removal will be obtained through chart review. For all failed catheters, re-insertion attempt data will be tracked through the medical record. If the patient is discharged prior to the time of follow-up assessment then the time of discharge will be documented and the VAD will be presumed functional until time of discharge unless otherwise noted in the chart. Some patients may leave the hospital with VAD in place for additional intravenous therapies. This information will be noted, but these patients will not receive follow-up assessments post-discharge for the research.If the patient has the midline longer than 7 days, the status of the line will be assessed via documentation in the electronic health record (EHR). The decision to remove the CVC is up to the treating physician.

Midline catheters will be assessed by research staff daily for usage. The medication administration record will be queried for all medications given through each catheter. Specifically, at the bedside we will assess whether the midline catheter is being used for any purpose. Of interest is the use of vesicants through the midline, medications that are generally given via central line or considered caustic to the vessel will be noted in both groups. Number of doses will be recorded.

Rates of symptomatic upper extremity superficial venous thrombosis (SVT) and deep venous thrombosis (DVT) rates, as confirmed by sonography will be calculated. Radiology interpretations will be reviewed for findings consistent with catheter-related symptomatic upper extremity venous thrombosis (CR-UEVT). This review will occur thirty days post patient discharge. Symptoms and rationale for imaging will be documented. If the patient is diagnosed with thrombophlebitis, the location of the thrombus will also be documented.

Infection rate will be tracked using confirmed catheter-related blood stream infection data from the surveillance team within the epidemiology department. The team utilizes the CDC definition of laboratory-confirmed blood-stream infection (LCBSI). The IV team will assess all IV insertions sites for infection.

The control data was collected as a separate IRB-approved study. Additional data for control and intervention groups includes but is not limited to: patient medical record number (MRN), sex, age, admission diagnosis (top 2), discharge diagnosis (top 2), admission from Emergency center/floor/transfer, Charlson Comorbidity Index (CCI), date of central line placement, date of central line removal, location of central line, number of lumens, medications with particular attention to drips and vesicants, ICU length of stay, hospital length of stay, disposition from the ICU, CLABSI. Baseline variables will be evaluated for differences between cases and controls. Matching will be used to select the controls used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older admitted to the MICU at Beaumont Hospital- Royal Oak who require a CVC Midline placement by the vascular access team within 24 hours of CVC placement

Exclusion Criteria:

* Patients not admitted to MICU
* Patients < 18 years of age
* Patients identified to require a PICC for extended duration of therapy
* Patients with midline catheters, pre-existing ports, dialysis catheters (Quinton), or other vascular access already inserted within the first 24 hours of CVC insertion (peripheral IV catheters are allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
CVC hours | at CVC removal, at any time up to 30 days
  Number of hours from CVC insertion to CVC removal

SECONDARY OUTCOMES:
CLABSI | 30 days
  Number of participants with catheter-related lab-confirmed blood stream infection per Center of Disease Control (CDC) guidelines
Upper extremity venous thrombosis | 30 days
  Number of participants with proven sonographic diagnosis of upper extremity deep vein thrombosis or superficial vein thrombosis
Midline IV catheter survival | 30 days
  Number of participants with midline catheter survival, defined as ability to withdraw 3-5 mls blood or flush without resistance with 5 ml saline daily, until completion of therapy
Midline Catheter Associated Phlebitis | 30 days
  Number of participants with each grade of phlebitis as assessed 0-5 Visual Phlebitis scale, where 0 indicates no phlebitis and 5 indicates advanced stages of thrombophlebitis

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No